CLINICAL TRIAL: NCT04078139
Title: Effects of Pre-emptive Scalp Infiltration With Ropivacaine and Methylprednisolone- Ropivacaine on Pain After Craniotomy in Adults
Brief Title: Pre-emptive Scalp Infiltration With Methylprednisolone Plus Ropivacaine for Postoperative Pain After Craniotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY 2018-034-02-5
Record Dates: First submitted 2019-09-02; First posted 2019-09-04 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Pain, Postoperative
Keywords: Postoperative Pain;; Post-Craniotomy;; Methylprednisolone; Ropivacaine; Scalp Infiltration
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The MP/RP group (Experimental): Participates will receive peri-incisional scalp infiltration with 10ml ropivacaine 1% wt/vol, 40mg methylprednisolone, plus 10ml saline;
  Interventions: Drug: The MP/RP group
- The RP group (Active Comparator): Participates will receive peri-incisional scalp infiltration with 10ml ropivacaine 1% wt/vol, plus 10ml saline;
  Interventions: Drug: The RP group

INTERVENTIONS:
Drug: The MP/RP group — Miscible liquid of methylprednisolone and ropivacaine in this study will be peri-incisional scalp infiltration with 40mg methylprednisolone, 10 ml 1% ropivacaine and 10 ml normal saline miscible liquids for participants who will undergo elective craniotomy. The local infiltration solution containing will be infiltrated along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigator.
  Arms: The MP/RP group
Drug: The RP group — Miscible liquid of ropivacaine in this study will be peri-incisional scalp infiltration with 10 ml 1% ropivacaine and 10 ml normal saline miscible liquids for participants who will undergo elective craniotomy. The local infiltration solution containing will be infiltrated along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigator.
  Arms: The RP group

SUMMARY:
Pain is common for the first 2 days after major craniotomy. A majority of patients would suffer from moderate-to-severe postoperative pain after undergoing craniotomy. Inadequate analgesia induced sympathetically mediated hypertension may lead to an increased risk for post-operative complications. Adequate pain control is essential for patients' prognosis and their postoperative life quality. Pain after craniotomy derives from the scalp and pericranial muscles. Local anesthetics administered around the incision have been performed clinically. However, some studies revealed that the analgesic effect of local anesthetics was not unsatisfactory due to its short pain relief duration. Pain is common for the first 2 days after major elective intracranial surgery, and the relatively short analgesic time of scalp infiltration does not seem to meet the requirements of craniotomy. Steroid such as methylprednisolone as an adjuvant to local anesthetics intra-articular injected locally reduced pain intensity after total knee arthroplasty or lumbar discectomy. However, there has not been reported about local application of methylprednisolone on scalp infiltration. Thus, the investigators suppose that pre-emptive scalp infiltration with steroid (methylprednisolone) plus local anesthetic (ropivacaine) could relieve postoperative pain after craniotomy in adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective craniotomy for resection of tumour under general anaesthesia;
* American Society of Anesthesiologists (ASA) physical status of I , II or III;
* Participates with an anticipated fully recovery within 2 hours postoperatively.

Exclusion Criteria:

* History of craniotomy;
* Expected delayed extubation or no plan to extubate;
* Participants who cannot use a patient-controlled analgesia (PCA) device;
* • Participants who cannot understand the instructions of a numeral rating scale (NRS) 35 before surgery;
* Extreme body mass index (BMI) (< 15 or > 35);
* Allergy to opioids, methylprednisolone or ropivacaine;
* History of excessive alcohol or drug abuse, chronic opioid use (more than 2 weeks), or use of drugs with confirmed or suspected sedative or analgesic effects;
* History of psychiatric disorders, uncontrolled epilepsy or chronic headache;
* Pregnant or at breastfeeding;
* Symptomatic cardiopulmonary, renal, or liver dysfunction or history of diabetes;
* Preoperative Glasgow Coma Scale< 15;
* Suspicion of intracranial hypertension;
* Peri-incisional infection;
* Participants who have received radiation therapy and chemotherapy preoperatively or with a high probability to require a postoperative radiation therapy and chemotherapy according to the preoperative imaging.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Estimated)
Dates: Start 2021-03-05 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative butorphanol consumption within 48 hours postoperatively | Within 48 hours after the operation
  All participates will receive an electronic intravenous patient-controlled analgesia (PCA) device. Participates will be advised to push the analgesic demand button if they feel pain.

SECONDARY OUTCOMES:
The number of participants who have no butorphanol consumption | Within 48 hours after the operation
  The number of participants who have not pushed the button of patient-controlled analgesia pump.
The first time to press the patient-controlled analgesia button | Within 48 hours after the operation
  The first time that the participants press the patient-controlled analgesia button.
The total times that participants press patient-controlled analgesia button | Within 48 hours postoperatively
  The total times that participants press patient-controlled analgesia button including effective presses and ineffective presses.
Numerical rating scale (NRS) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months and 6 months after surgery
  Pain will be assessed after surgery by numerical rating scale (0 indicates no pain, 10 indicates the most severe pain imaginable).
Postoperative nausea and vomiting | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Postoperative nausea and vomiting (PONV) was rated by participates as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; and 3, vomiting.
Ramsay Sedation Scale (RSS) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Ramsey 1: Anxious, agitated, restless; Ramsey 2: Cooperative, oriented, tranquil; Ramsey 3: Responsive to commands only If Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.
Respiratory depression | Within 48 hours after the operation
  Respiratory depression is defined as a respiratory rate less than 10 breaths per minute or oxygen saturation was less than ninety percent.
The times of emergency reducing blood pressure after the operation | Within 48 hours after the operation
  The criteria for treatment is determined by the participant's surgeon in charge.The times of emergency reducing blood pressure will be recording by the investigator.
Patient satisfactory scale (PSS) | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months and 6 months after surgery
  0 for unsatisfactory, and 10 for very satisfied
The total consumption of opioids during the operation | During procedure
  The total consumption of opioids during the operation
The length of stay | Approximately 2 weeks after the surgery
  The duration of hospitalization after the operation
The World Health Organization Quality of Life (WHOQOL)-BREF | At 1 month, 3 months and 6 months after surgery
  Quality of life will be measured using the World Health Organisation QoL-BREF (WHOQOL-BREF) questionnaire. The WHOQOL-BREF is a abbreviated version of the WHOQOL-100 assessment. WHOQOL-BREF is a self-report questionnaire that contains 26 items and addresses 4 QOL domains: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). Two other items measure overall QOL and general health. Each domain's mean score can range between 4 and 20 and a higher score indicates a higher quality of life. The mean score of items within each domain is used to calculate the domain score. A transformation method converts domain scores to a 0-100 scale.
Wound Healing Score | At 1 month after surgery
  Skin Healing 1: fully healed; 2: ≤3 cm in total not healed; 3: >3 cm not healed; 4: areas of necrosis ≤3 cm; 5: areas of necrosis >3 cm Infection 1: none; 2: ≤0.5-cm margin of redness; 3: more redness or superficial pus; 4: deep infection; not applicable Hair Regrowth 1: even regrowth along wound; 2: ≤3 cm not regrowing; 3: >3-6 cm not regrowing; 4: >6 cm not regrowing; not applicable

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gurbet A, Bekar A, Bilgin H, Ozdemir N, Kuytu T. Preemptive wound infiltration in lumbar laminectomy for postoperative pain: comparison of bupivacaine and levobupivacaine. Turk Neurosurg. 2014;24(1):48-53. doi: 10.5137/1019-5149.JTN.8431-13.0. PMID 24535791
- [Background] Ersayli DT, Gurbet A, Bekar A, Uckunkaya N, Bilgin H. Effects of perioperatively administered bupivacaine and bupivacaine-methylprednisolone on pain after lumbar discectomy. Spine (Phila Pa 1976). 2006 Sep 1;31(19):2221-6. doi: 10.1097/01.brs.0000232801.19965.a0. PMID 16946657
- [Background] Mullaji A, Kanna R, Shetty GM, Chavda V, Singh DP. Efficacy of periarticular injection of bupivacaine, fentanyl, and methylprednisolone in total knee arthroplasty:a prospective, randomized trial. J Arthroplasty. 2010 Sep;25(6):851-7. doi: 10.1016/j.arth.2009.09.007. Epub 2009 Dec 21. PMID 20022457
- [Background] Rocha-Filho PA. Post-craniotomy headache: a clinical view with a focus on the persistent form. Headache. 2015 May;55(5):733-8. doi: 10.1111/head.12563. Epub 2015 Apr 22. PMID 25903913
- [Background] Tsaousi GG, Logan SW, Bilotta F. Postoperative Pain Control Following Craniotomy: A Systematic Review of Recent Clinical Literature. Pain Pract. 2017 Sep;17(7):968-981. doi: 10.1111/papr.12548. Epub 2017 Feb 23. PMID 27996204
- [Background] Dunn LK, Naik BI, Nemergut EC, Durieux ME. Post-Craniotomy Pain Management: Beyond Opioids. Curr Neurol Neurosci Rep. 2016 Oct;16(10):93. doi: 10.1007/s11910-016-0693-y. PMID 27604271
- [Background] Rahimi SY, Alleyne CH, Vernier E, Witcher MR, Vender JR. Postoperative pain management with tramadol after craniotomy: evaluation and cost analysis. J Neurosurg. 2010 Feb;112(2):268-72. doi: 10.3171/2008.9.17689. PMID 19630495